CLINICAL TRIAL: NCT05731076
Title: Efficacy of Self-Management Support on Nutritional Status in Lung Cancer Patients With Cancer Cachexia Syndrome: A Randomized Clinical Trail
Brief Title: Self-Management Support for Lung Cancer Patients With Cachexia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Chang Li Chun, Head of nurse practitioner, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 220582
Record Dates: First submitted 2023-01-23; First posted 2023-02-16 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Cachexia-Anorexia Syndrome
Keywords: cancer cachexia syndrome; exercise; nutrition; muscle endurance; body mass index
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management support nutrition and exercise group (Experimental): Educate how to plain regular exercise and eat enough protein diet with self-management support.
  Interventions: Behavioral: Self-management support nutrition and exercise intervention
- Routine health education group (No Intervention): Routine health education.

INTERVENTIONS:
Behavioral: Self-management support nutrition and exercise intervention — Provide information about different home exercise type(walking, strength training, flexibility training), nutrition knowledge to maintain or improve cancer cachexia syndrome.
  Arms: Self-management support nutrition and exercise group

SUMMARY:
The goal of this randomized clinical trial is to test the efficacy of self-management support based exercise combine nutrition intervention in lung cancer patient with cancer cachexia anorexia syndrome . The main question it aims to answer is:

• Would exercise combine nutrition intervention improve lung cancer patients' nutrition status? Participants will make custom exercise plan and eat enough protein food after self-management support based education.

And there is a comparison group: Researchers will compare comparison group to see nutrition status who receive routine health education.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed lung cancer(ICD-10 code: C33-C34)
2. Body weight loss: body weight loss 2% before recruitment 2 months or body weight loss 5% before recruitment 6months.
3. Physician judged may do home exercise without supervisor.
4. Has smart phone and agree to use exercise associated application.
5. Agree to wear Xioami smart band as long as passible.
6. Conscious clear and communication.
7. Eastern Cooperative Oncology Group (ECOG) 0-1.

Exclusion Criteria:

1. Participants with cardiovascular disease can't exercise without supervisor.
2. Diabetes Mellitus with blood sugar poor control.
3. Chronic obstructive pulmonary disease with dyspnea on exertion.
4. Platelets < 50000mm3 due to disease or treatment.
5. Hemoglobin <10mg/dl.
6. Recently stumble, severe pain, cognitive and behavior change.
7. Suspect or diagnosed brain metastasis.
8. Suspect or diagnosed bone metastasis.
9. Receive Nasogastric tube feeding or parenteral nutrition.
10. Physician judged can't do home exercise.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change form Minimal Nutrition Assessment(MNA) at 12 weeks | Before allocation and after intervention 8 and 12 weeks.
  The MNA consists of 18 self- reported questions. Each question has different score and marked near the answer. The first part of MNA is six questions about ingestion, weight loss, current mobility, an acute illness or major stress, a neuropsychological problem, and a decrease in body mass index. The second part evaluates living arrangements, the presence of polypharmacy or pressure ulcers, the number of full meals eaten daily, the amount and frequency of specific foods and fluids, and the mode of feeding. The patient reports nutritional and health status, and the practitioner determines weight and height (to calculate BMI), and mid-arm and mid-calf circumferences. The maximal score is 30, score >23.5 means well-nourished, 17~23.5 means risk of malnutrition, < 17 means malnutrition.
Change from body weight at 12weeks | Before allocation and after intervention 8 and 12 weeks.
  The body wight will be detected by OMRON HBF-375. Data record in kilograms and after the first decimal place.
Change from body fat mass at 12weeks | Before allocation and after intervention 8 and 12 weeks.
  The body fat mass will be detected by OMRON HBF-375. Data record with percentage and after the first decimal place.
Change from muscle mass at 12weeks | Before allocation and after intervention 8 and 12 weeks.
  The muscle mass will be detected by OMRON HBF-375. Data record with percentage and after the first decimal place.

SECONDARY OUTCOMES:
30 second arm curl test | Before allocation and after intervention 8 and 12 weeks.
  Used to test muscle endurance of upper extremities. Let the participant sit on a chair and holding the dumbbell(female 5 pound; male 8 pound), then repeated curl his/her elbow. Count how many times can the participant curl their elbow in 30 seconds. More curl times means better upper endurance.
30 second chair-stand test | Before allocation and after intervention 8 and 12 weeks.
  To test muscle endurance of lower extremities. Let the participant sit on a chair, then repeated stand up and sit. Count how many times can he/she curl his/ her elbow in 30 seconds. The more frequency the better lower limb endurance.
Six-minute walking test | Before allocation and after intervention 8 and 12 weeks.
  Examine cardiopulmonary function in this study. Let the participant sit and rest 10 minutes before test. Check vital signs and oxygen situation for patient safety. Position the participant at the starting line, and walking back and forth along the mark on the floor. When the participant starts to walk, starts the times. Don't walk nor talk with him/ her, and count the laps attentively. Participant can walk longer distance means better cardiopulmonary function.
Functional Assessment of Cancer Therapy- Lung (FACT-L) | Before allocation and after intervention 12 weeks.
  FACT-L could determine quality of life in lung cancer patients. It content 5 dimensions, physical well-being 7items, social/family well-being 7items, emotional well-being 6items, functional well-being 7 items, and Lung cancer sub-scale 9 items. It used Likert 5 point and the score ranged from 0 to 144. The higher score means better quality of life.
Cancer anorexia-cachexia syndrome nutrition knowledge scale | Before allocation and after intervention 12 weeks.
  Cancer anorexia-cachexia syndrome nutrition knowledge scale was developed to test cancer patients' cachexia nutrition knowledge. It content the knowing of cancer anorexia-cachexia syndrome(7 items), the technology on choose food(15 items), and anorexia management(7 items). The items are multiple choice but only one correct answer. The score ranged from 0 to 29, the higher score means the participant has better nutrition knowledge to against cancer anorexia-cachexia syndrome.
24 hours dietary recall | Before allocation and after intervention 8 and 12 weeks.
  To understand participants' nutrition intake before and after intervention. Let participants recall their last 24 hours diet by interview, include dish name, amount, cooking method, and nutrition supply. Collected data will be translated to calories, protein, fat, and carbohydrate by a nutritionist, and then it will be continues variable for analysis.
Change from amount of exercise at 12 weeks | Collect 1~8week and 8-12 week exercise record.
  Measure amount of exercise by Xioami smart band. It is a wearable device, can record exercise, include time, duration, and heart rate...etc. Let the participant wear the smart band all day if passible. Collect walking distance, exercise date, exercise mode, duration by latest Xioami published application. Collected data will be continuous variable and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Li Chun Chang, Master, Principal Investigator — Yuanlin Christian hospital
Locations (2):
- Taiwan (2):
  - Yuanlin Christian Hospital, Changhua
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615
- [Background] Anderson LJ, Albrecht ED, Garcia JM. Update on Management of Cancer-Related Cachexia. Curr Oncol Rep. 2017 Jan;19(1):3. doi: 10.1007/s11912-017-0562-0. PMID 28138933
- [Background] Ozaki H, Nakagata T, Yoshihara T, Kitada T, Natsume T, Ishihara Y, Deng P, Kobayashi H, Machida S, Naito H. Effects of Progressive Walking and Stair-Climbing Training Program on Muscle Size and Strength of the Lower Body in Untrained Older Adults. J Sports Sci Med. 2019 Nov 19;18(4):722-728. eCollection 2019 Dec. PMID 31827357
- [Result] Muscaritoli M, Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Oldervoll L, Ravasco P, Solheim TS, Strasser F, de van der Schueren M, Preiser JC, Bischoff SC. ESPEN practical guideline: Clinical Nutrition in cancer. Clin Nutr. 2021 May;40(5):2898-2913. doi: 10.1016/j.clnu.2021.02.005. Epub 2021 Mar 15. PMID 33946039
- [Result] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Result] Peddle-McIntyre CJ, Singh F, Thomas R, Newton RU, Galvao DA, Cavalheri V. Exercise training for advanced lung cancer. Cochrane Database Syst Rev. 2019 Feb 11;2(2):CD012685. doi: 10.1002/14651858.CD012685.pub2. PMID 30741408
- [Result] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Result] Schreiber M, Bucher T, Collins CE, Dohle S. The Multiple Food Test: Development and validation of a new tool to measure food choice and applied nutrition knowledge. Appetite. 2020 Jul 1;150:104647. doi: 10.1016/j.appet.2020.104647. Epub 2020 Feb 29. PMID 32119883